CLINICAL TRIAL: NCT07060729
Title: Exploring How Exercise Frequency Impacts Muscle Resistance and Balance in Institutionalized Seniors: Protocol for a Randomized Controlled Trial
Brief Title: Exploring How Exercise Frequency Impacts Muscle Resistance and Balance in Institutionalized Seniors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Leiria (Other)
Responsible Party: Principal Investigator, Filipe Fernandes Rodrigues, Doctorate, Instituto Politécnico de Leiria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IPLEIRIA/59/2022
Record Dates: First submitted 2025-06-23; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Frequency of Treatment Protocol
Keywords: Institutionalization; Frequency; Exercise; Fall risk; Muscle strength
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral: 2 exercise sessions (2X) (Active Comparator): The (1) control group (2X) will receive an exercise screening checklist and 24 group training sessions, 2 times per week during a 12-week period, based on International Exercise Recommendations in Older Adults (ICFSR; Izquierdo et al., 2021). These are the recommendations commonly used for older adults.
  Interventions: Behavioral: Behavioral: 2 exercise sessions (2X)
- Behavioral: 3 exercise sessions (3X) (Experimental): The (3) experimental group (3X) will receive an exercise screening checklist and 36 group training sessions, 3 times per week during a 12-week period, based on International Exercise Recommendations in Older Adults (ICFSR; Izquierdo et al., 2021). These are the recommendations commonly used for older adults. This additional session will increase weekly exercise volume compared to the control group, also being closer to complying to the WHO International Guidelines of weekly physical activity (Bull et al., 2020)
  Interventions: Behavioral: Behavioral: 2 exercise sessions (3X)

INTERVENTIONS:
Behavioral: Behavioral: 2 exercise sessions (2X) — The (1) control group (2X) will receive an exercise screening checklist and 24 group training sessions, 2 times per week during a 12-week period, based on International Exercise Recommendations in Older Adults (ICFSR; Izquierdo et al., 2021). These are the recommendations commonly used for older adults.
  Arms: Behavioral: 2 exercise sessions (2X)
Behavioral: Behavioral: 2 exercise sessions (3X) — The (3) experimental group (3X) will receive an exercise screening checklist and 36 group training sessions, 3 times per week during a 12-week period, based on International Exercise Recommendations in Older Adults (ICFSR; Izquierdo et al., 2021). These are the recommendations commonly used for older adults. This additional session will increase weekly exercise volume compared to the control group, also being closer to complying to the WHO International Guidelines of weekly physical activity (Bull et al., 2020)
  Arms: Behavioral: 3 exercise sessions (3X)

SUMMARY:
The older population is the least likely to engage in regular physical activity and to meet international recommendations for performing 150 minutes of moderate-intensity physical activity per week. Additionally, older adults living in care institutions tend to have even lower levels of physical activity compared to those living in the community. This physical inactivity among institutionalized older adults carries harmful consequences, such as the loss of muscle mass and strength, both of which are associated with decreased balance and an increased risk of falling, an adverse event with personal, physical, economic, social, and potentially fatal implications. Although this situation is well described in the literature, little is known about whether increasing physical activity levels from near-optimal (almost 150 minutes of physical activity per week) to optimal (more than 150 minutes per week) can influence muscle strength and balance in institutionalized older adults, and thereby reduce the burden related to falls.

This type of research is essential, as weekly frequency may be a variable to consider in the prescription of physical exercise for this population. The American College of Sports Medicine (ACSM) recommends using the FITT principle (Frequency, Intensity, Type, and Time) to guide exercise prescription. By adjusting these factors, individuals can tailor workouts to their specific goals and fitness levels. While attention has been given to the type of training, its intensity, and its duration, it is important to recognize that total weekly volume may be a determining factor for improvements in components of physical fitness.

Considering that this population tends to be physically inactive, incorporating physical activity two or three times per week may lead to different outcomes. While exercising twice per week may seem suboptimal, as it does not meet international guidelines, engaging in physical activity three times per week may be the minimum necessary to observe positive effects on muscle strength and balance.

DETAILED DESCRIPTION:
Ageing is a universal experience. However, the physical ageing process occurs differently across individuals. When individuals remain physically active throughout life, their levels of physical fitness tend to be higher compared to those with low or no engagement in physical activity. Nevertheless, the literature shows that the general population does not meet the international recommendation of 150 minutes of moderate-intensity physical activity per week, and that the proportion of physically inactive individuals is higher among the older population compared to adults or children.

Given this scenario, marked by a lack of physical activity and the gradual loss of muscle mass inherent to ageing, which is exacerbated by the absence of muscular and cardiovascular stimulation, there is an increased risk of adverse outcomes, such as falls. It is well documented in the literature that physically inactive ageing is more pronounced in older adults living in institutions compared to those who remain in the community. This may be because community-dwelling older adults typically engage in behaviors considered physically active, such as household chores, social and recreational activities outside the home, gardening, or do-it-yourself tasks that promote movement. Conversely, older adults in institutional care, who are typically institutionalized due to a lack of autonomy and independence, tend to experience an accelerated physical ageing process, given the general lack of opportunities for physical activity. In such settings, household chores are not typically performed, opportunities to leave the premises for social or recreational activities are limited, and access to gardening spaces is often unavailable. Thus, institutionalized older adults are more vulnerable to the effects of physical inactivity, which further increases dependency on others.

The literature consistently highlights the beneficial effects of physical activity on the quality of life of older adults, including those living in institutions. Reducing the risk of falling is essential, as such events may result in total dependence, such as becoming bedridden or reliant on a wheelchair, and often involve a longer and more demanding recovery, both physically and psychologically. Falls also incur various costs: individual (e.g., medication), public (e.g., medical treatments), and institutional (e.g., hiring additional staff). Furthermore, fear of engaging in physically active behaviors, such as walking, due to the potential risk of falling again, can further discourage movement. Understanding that physical activity can play a protective role, by reducing fall risk, increasing confidence in physical activity, and gradually promoting independence and autonomy, may yield benefits both for the individual and for all parties involved in the care of institutionalized older adults.

In terms of international recommendations, the World Health Organization (WHO) and the American College of Sports Medicine (ACSM) advise that individuals perform at least 150 minutes of moderate-intensity physical activity per week, preferably 30 minutes per day. Additionally, strength training is recommended at least twice per week, at moderate intensity, involving 8-10 exercises and 10-15 repetitions per set. Flexibility and balance training are also advised twice per week, with each stretch lasting 15-30 seconds and repeated 2-4 times per muscle group, using static, dynamic, passive, or active exercises. However, despite being labelled as "recommendations," these guidelines present several practical limitations for the institutionalized older population. First, they imply approximately 60-90 minutes of regular physical activity per day, a significantly high volume for a population that is, by nature, physically inactive. Second, transitioning from inactivity to 60-90 minutes of daily exercise may be too abrupt, especially in the absence of appropriate adaptation and progression, and may increase the risk of adverse events associated with existing metabolic or cardiovascular conditions. Third, according to the ACSM, institutionalized older adults already present with at least one (or more) cardiovascular risk factor, requiring more cautious approaches than those applied to community-dwelling older adults or younger individuals. Lastly, not all institutions have access to resistance or cardio machines, free weights, transport to fitness facilities, or supervised professional guidance, which may limit the implementation of the strength training recommended by the WHO and ACSM.

Given this context, physical activity prescription for this population requires a tailored methodology suited to the institutional setting, namely, through multicomponent exercise programs. These programs integrate various components of physical fitness, including cardiovascular endurance, muscular strength, balance, agility, and flexibility. Sessions typically last 45-60 minutes and are conducted at light to moderate intensity, individualized based on each participant's subjective perception of effort, thereby allowing for self-regulation of intensity according to individual capabilities. According to the FITT framework, three of the four principles (Intensity, Type, and Time) are thereby addressed, with Frequency remaining as the variable to be further explored.

The variable of frequency is considered essential, as it can be pragmatically adjusted for populations residing in institutional settings. Multicomponent programs have traditionally been implemented two or three times per week, with a rest interval of one to two days between sessions. This schedule facilitates a cycle of physical stimulation followed by recovery. Furthermore, participation in two or three sessions per week, each lasting 45-60 minutes, presents a noteworthy distinction: two sessions fall short of the 150-minute weekly recommendation, while three sessions slightly exceed this threshold. Nevertheless, participation in such programs two or three times per week has demonstrated significant benefits across multiple domains of physical fitness, including cardiovascular endurance, muscular strength, balance, and agility. Thus, even without strict compliance with existing recommendations, substantial benefits are evident. The aim of the present investigation is to determine whether increased frequency yields greater benefits in this population, and whether greater emphasis should be placed not on rigid thresholds (e.g., the 150-minute guideline), but rather on identifying the minimum effective dose required to transition physically inactive institutionalized older adults to an "active" status during the initial stages of engagement in a multicomponent exercise program. The findings may support professionals in tailoring interventions to increase muscle mass and reduce fall risk among institutionalized older adults.

ELIGIBILITY:
Inclusion criteria:

* 65 years to 90 years.
* Apparently healthy and without medical contraindications to exercise.
* Normal weight (BMI ≤ 24.99 kg/m2) or overweight (BMI > 25 ≤ 29.99 kg/m2)
* Being institutionalized for more than 6 months.
* Not having done any exercise regime for the last 6 months or any kind of structured sport activity.

Exclusion criteria

Before Enrollment:

* High risk of cardiovascular disease (ACSM, 2021)
* High blood pressure (≥ 140/90mmHg) in the pre-exercise evaluation (ESC, 2024)
* High risk of fall (more than 1 fall over the last 6 months).

During the intervention:

* Acquired injury.
* Acquired medical condition.
* Related or not related fall during intervention.
* Inability to perform 5 consecutive exercise sessions.
* Exercise adherence below 75% of total sessions (n = 24 or n = 36)

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Training sessions attendance rate | Baseline and at week 13 (after 12 week of intervention)
  Post-intervention weekly exercise frequency, objectively measured by the physiologist using an attendance sheet.

SECONDARY OUTCOMES:
Waist measurement | Baseline and at week 13 (after 12 week of intervention)
  Waist measurement is determined by using the midpoint between the lowest rib and the top of the hip bone, then wrapping a measurement tape around the waist.
Height | Before intervention
  Height is determined by the vertical distance of the person from the base to the top using a stadiometer.
Weight | Baseline and at week 13 (after 12 week of intervention)
  Weight is determined by the body mass of a person on a calibrated scale.
Body Mass Index | Baseline and at week 13 (after 12 week of intervention)
  Body Mass Index is calculated by dividing weight in kilograms by the square of height in meters.
Balance and dynamic agility measured using the Timed Up and Go test | Baseline and at week 13 (after 12 week of intervention)
  Timed up and Go is measured by timing how long it takes a person to stand up from a chair, walk 2.44 meters, turn around, walk back to the chair, and sit down.
Upper body muscle resistance measured using the Arm curl test | Baseline and at week 13 (after 12 week of intervention)
  Arm curl test is measured by assessing how many bicep curls using a dumbbell (4-5 lbs for women, 8 lbs for men) a person can complete in 30 seconds
Lower body muscle resistance measured using the Chair sit and stand test | Baseline and at week 13 (after 12 week of intervention)
  Chair sit and stand test is measured by counting the number of sit-to-stand repetitions completed within 30 seconds.
Rate of Falls per participant | Baseline and at week 13 (after 12 week of intervention)
  Reported by the physiologists or by medical and nursing staff within the institution.

OTHER OUTCOMES:
Resting blood pressure (mmHg) | Before training session
  Resting blood pressure is measured using an arm sleeve equipment monitor by placing the cuff so that its lower edge is about three centimeters above the elbow and the arm is supported on a table, so that the cuff is at the level of your heart.
Resting heart rate before exercise (bpm) | Before training session
  Resting heart rate is measured using an arm sleeve equipment monitor by placing the cuff so that its lower edge is about three centimeters above the elbow and the arm is supported on a table, so that the cuff is at the level of your heart.
Exercise intensity | After 10, 30, and 60 minutes of each training session, and data reported will be light (1 point), moderate (2 points) or vigorous intensity (3 points).
  Exercise intensity is measured using the talk test, which considers the ability a person can talk and/or breathe and based on that, determined intensity.

IPD SHARING:
Plan to Share IPD: Yes
Primary and secondary data related to the study.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After publication.
Access Criteria: University teachers and reseachers.

REFERENCES:
- [Background] Rodrigues F, Izquierdo M, Monteiro D, Jacinto M, Matos R, Amaro N, Antunes R, Teixeira DS. Muscle Strength Matters Most for Risk of Falling Apart from Body Mass Index in Older Adults: A Mediated-Moderation Analysis. J Frailty Aging. 2024;13(4):427-431. doi: 10.14283/jfa.2024.68. PMID 39574263
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Background] Izquierdo M, Merchant RA, Morley JE, Anker SD, Aprahamian I, Arai H, Aubertin-Leheudre M, Bernabei R, Cadore EL, Cesari M, Chen LK, de Souto Barreto P, Duque G, Ferrucci L, Fielding RA, Garcia-Hermoso A, Gutierrez-Robledo LM, Harridge SDR, Kirk B, Kritchevsky S, Landi F, Lazarus N, Martin FC, Marzetti E, Pahor M, Ramirez-Velez R, Rodriguez-Manas L, Rolland Y, Ruiz JG, Theou O, Villareal DT, Waters DL, Won Won C, Woo J, Vellas B, Fiatarone Singh M. International Exercise Recommendations in Older Adults (ICFSR): Expert Consensus Guidelines. J Nutr Health Aging. 2021;25(7):824-853. doi: 10.1007/s12603-021-1665-8. PMID 34409961
- [Background] Mollinedo Cardalda I, Lopez A, Cancela Carral JM. The effects of different types of physical exercise on physical and cognitive function in frail institutionalized older adults with mild to moderate cognitive impairment. A randomized controlled trial. Arch Gerontol Geriatr. 2019 Jul-Aug;83:223-230. doi: 10.1016/j.archger.2019.05.003. Epub 2019 May 8. PMID 31100545